CLINICAL TRIAL: NCT01306370
Title: Prevention of Postoperative Blood Loss: Randomised Unicentric Parallel Clinical Trial That Assess the Efficacy of Fibrin Glue and Tranexamic Acid in Surgical Patients With a Total Knee Arthroplasty.
Brief Title: Fibrin Glue or Tranexamic Acid for Total Knee Arthroplasty
Acronym: ATRHEMOS
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Collaborators: Banc de Sang i Teixits (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 2009-017804-95; TRA-81 (Other Grant/Funding Number: Spanish Health Ministry and Social Policy)
Record Dates: First submitted 2011-02-28; First posted 2011-03-01 (Estimated); Last update posted 2013-08-28 (Estimated); Status verified 2013-08

CONDITIONS: Knee Arthropathy
Keywords: primary knee arthroplasty; fibrin glue; tranexamic acid; topic
MeSH Terms: interventions — Tranexamic Acid; Fibrin Tissue Adhesive

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (4):
- Tranexamic acid (Experimental): Tranexamic acid is a synthetic derivative of the amino acid lysine. It inhibits fibrinolysis by blocking the lysine binding sites on plasminogen and facilitates the coagulation process.
  Interventions: Drug: Tranexamic Acid
- Fibrin glue BSTC (Experimental): It is homologous fibrin glue from a single blood donor.
  Interventions: Biological: Fibrin glue
- Tissucol (Experimental): It is fibrin glue commercialized from multiple donors.
  Interventions: Drug: Fibrin glue
- Habitual haemostasis (Other): Electrocoagulation of blood vessels was performed during surgery in all patients (routine hemostasis)
  Interventions: Other: Habitual haemostasis

INTERVENTIONS:
Drug: Tranexamic Acid — Two dosage during the surgical intervention: the first dosage 15-30' before the leg ischemia and the second dosage at 60 -90' after the first dosage.
  Each dosage: 2 ampoules of 500mg/5 mL/ampoule
  Other Names: Amchafibrin
  Arms: Tranexamic acid
Drug: Fibrin glue — Topical administration, before to close the surgical wound. Dosage: 2 mL.
  Other Names: Tissucol
  Arms: Tissucol
Biological: Fibrin glue — Topical administration, before to close the surgical wound.
  Arms: Fibrin glue BSTC
Other: Habitual haemostasis — The surgical habitual haemostasis.
  Arms: Habitual haemostasis

SUMMARY:
Objectives:

a) Principal: To assess if the fibrin glue or the tranexamic acid reduce less than 20% the blood losses with respect to the habitual haemostasia in patients with arthroplasty total of knee.

Secondaries: To assess the treatment safety. To perform a cost- analyses.

Methods: Randomized, unicentric, and parallel clinical trial with four comparative groups: Tissucol® (fibrin glue), fibrin glue manufactured by the Cryoseal® system (Banc de Sang i Teixits de Catalunya), tranexamic acid and habitual haemostasia.

Nº of participant centres: 1. Random allocation will be centralised.

Main outcome: Blood losses (ml) in the post-operatory period collected by the habitual drain system.

Secondary outcomes: Proportion of patients with blood transfusion, complications of surgery wound, pre and post-operative haemoglobin, units of blood transfused, post-operative mortality, days of hospital stay, safety of interventions assessed.

Size sample calculation: The number needed of patients is 172 (43 per group) to demonstrate a 20% difference in the post-operative blood losses between the treatments assessed and the habitual haemostasia, with a statistical power of 80% and a 0.05 bilateral alpha, and a 20% of withdrawals.

Statistical analysis: The investigators will perform a comparison of outcomes through the "t" test, the Mann-Whitney test of chi square, depending of the evaluated outcomes, quantitative or ordinals or qualitative, respectively. The software used will be Statistical Package for the Social Sciences (SPSS) version 17.

ELIGIBILITY:
Inclusion Criteria:

* Total knee arthroplasty
* The patient consent to participate

Exclusion Criteria:

* Intolerance drugs to the study or to bovine protein (aprotinin)
* Antecedent of thromboembolic disease
* Patient with cardiac alterations of the rhythm
* Patients with valvular cardiac prosthesis
* Patients with pro-thrombotic alterations of coagulation
* Treatment with anticonceptive drugs

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 172 (Actual)
Dates: Start 2010-06; Primary Completion 2011-10 (Actual); Study Completion 2011-11 (Actual)

PRIMARY OUTCOMES:
Postoperative blood loss (mL) | During the first 48h after the surgical intervention
  Blood loss (mL) by the surgical wound collected by drain systems.

SECONDARY OUTCOMES:
Percentage of patients that need a postoperative blood transfusion | During the first postoperative week
Percentage of patients with surgical wound infection | During the first postoperative month
Percentage of patients with surgical wound dehiscence | During the first postoperative month
Percentage of patients with re-intervention by wound complications | During the first postoperative month
Incidence of deep venous thrombosis | During the first postoperative week
Pain of surgical wound | During the first postoperative week
Units of blood transfusion | During the first postoperative week
hospital length stay | Days
Mortality | During the first postoperative month

CONTACTS AND LOCATIONS:
Overall Officials: Martinez Zapata, Mª José, Study Director — Centro Cochrane Iberoamericano. Servicio de Epidemiología Clínica y Salud Pública. IIB Sant Pau; Aguilera Roig, Xavier, Principal Investigator — Hospital de la Santa Creu i Sant Pau. IIB Sant Pau
Locations (1):
- Hospital de la Santa Creu i Sant Pau, Barcelona, Catalonia, Spain